CLINICAL TRIAL: NCT04185298
Title: Mobile Technology-Based Simultaneous Aerobic Exercise and Memory Training Intervention for Older Adults With Mild Cognitive Impairment
Brief Title: mSIM: Mobile Simultaneous Aerobic Exercise and Memory Training Intervention for Amnestic Mild Cognitive Impairment
Acronym: mSIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in recruitment and completion rates, the study was considered to be not feasible. After 4 years, only 12 participants were randomized. Of the 8 mSIM arm participants, only 2 completed the study.
Sponsor: Jennifer Bramen (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Jennifer Bramen, Assistant Professor, Saint John's Cancer Institute
Organization: Saint John's Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191298; R21AG061494 (NIH)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Amnestic Mild Cognitive Impairment

STUDY DESIGN:
Intervention Model Description: The study will include two arms: Arm 1: activity monitoring only control (CON), Arm 2: active intervention with mSIM program (mSIM) plus activity monitoring (via Fitbit), to evaluate the efficacy of the mSIM intervention on memory performance and everyday functioning. The 'Activity monitoring only' arm will serve as the control group. Study objectives include measuring treatment related changes in memory performance and everyday functioning along with putative biomarkers of the behavioral changes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No treatment) (Active Comparator): Group 1: Participants will have continuous activity monitoring (via Fitbit)
  Interventions: Behavioral: mSIM intervention plus activity monitoring
- Group 2 (Experimental) (Experimental): Group 2: Participants will receive the mSIM treatment and have their activity monitored continuously (via Fitbit)
  Interventions: Behavioral: Activity monitoring

INTERVENTIONS:
Behavioral: mSIM intervention plus activity monitoring — Participants will receive the full mSIM intervention and be monitored (via Fitbit)
  Arms: Group 1 (No treatment)
Behavioral: Activity monitoring — Participants will have activity monitored (via Fitbit)
  Arms: Group 2 (Experimental)

SUMMARY:
The mSIM study involves developing and conducting feasibility testing of a web-based application that will deliver mobile-based simultaneous exercise and memory skills training program (mSIM) for amnesic Mild Cognitive Impairment (aMCI) patients.

The randomized control trial (RCT) will evaluate the efficacy of mSIM on memory performance and everyday functioning using 2 study arms (Group 1 activity monitoring control (via Fitbit) (CON) vs Group 2 mSIM intervention plus activity monitoring via Fitbit). mSIM treatment response will be evaluated using neuropsychological and functional evaluation. Concentration levels of peripheral biomarkers Brain-derived neurotrophic factor (BDNF) and norepinephrine (NE) also be assessed.

DETAILED DESCRIPTION:
The purpose of the study is to create a web-based cognitive compensatory, and predominately memory skills, training course that is delivered on a mobile device and compatible with use on a stationary bicycle and test its efficacy on memory and functional ability.

Participants will be recruited from (1) the Pacific Brain Health Center in Santa Monica, which is a high-volume memory-care and dementia outpatient clinic within a large physician medical group affiliated with Providence Saint John's Health Center, (2) advertisement to participants in the local community, and (3) establishment of a website landing page that permits interested individuals to contact the trial coordinator. Up to five participants will be course beta testers. They will receive a truncated version of the course and will provide detailed feedback. 30 participants will be randomized into one of two groups. Group 1 (control arm) will have their physical activity levels continuously monitored (via Fitbit). Participants will receive the Experimental Research Subject's Bill of Rights prior to signing the informed consent form (ICF), authorization of use and disclosure of protected health information (PHI), and authorization of medical record release for the subject's treating physician, will be obtained from each participant prior to enrolling in the study. A copy of all signed ICF's will be given to the participants, and the investigator will retain the original.

Group 2 (active arm) will receive the mSIM intervention plus activity monitoring (via Fitbit). Group 2 will first undergo 2-6 week of an exercise ramp-up (2x/week) until they can sustain 40 minutes at 50% heart rate reserve (HRR). The intensity for mSIM training will be 40-60% HRR. After the ramp-up phase the mSIM participants will begin the 12-week intervention, comprised of 2 60-minute sessions/week. mSIM treatment response will be evaluated using neuropsychological and functional evaluation. Assessments will occur at baseline, mid-trial (3-4 months) and post-trial (5-6 months). Concentration levels of peripheral biomarkers BDNF and NE at baseline and post-trial (5-6 months) will also be assessed.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be age 50 to 80 at time of informed consent.
* Subjects must confirm an aMCI diagnosis either by providing records from a clinical assessment within 6 months of enrollment in this study or through a brief memory assessment by study staff at screening.
* Subjects must be proficient in spoken and written English for consenting as well as for study participation since the intervention in this study is currently only available in English.
* Subjects with medical conditions must be stable for these conditions. Stable control on medication is acceptable.
* Subjects, with or without assistance, must be able to use a computer and web interface. If assistance is needed, it must be readily available to them.
* Subjects are required to have internet with Wi-Fi at the location of their mSIM training.
* Subject must have normal visual acuity (or corrected to normal) and normal color vision as indicated by self-report.
* Subject must have adequate hearing acuity as indicated by self-report.
* Subject must have adequate motor capacity to use a mobile phone/iPad/computer as indicated by self-report.
* Subjects must be able to provide medical clearance to participate in an unsupervised, moderate intensity exercise program from a physician.

Exclusion Criteria

* Subjects must not have an existing diagnosis of a neurodegenerative disorder (e.g., Alzheimer's Disease, Lewy Body Dementia, Frontal-Temporal Dementia).
* Subjects must not have a prior diagnosis that might impact cognition and movement abilities including: significant cardiovascular disease, significant respiratory disease, illness or injury, substance abuse, schizophrenia, bipolar disorder, or other neurological diseases.
* Subjects must not have a previous Mini Mental State Exam (MMSE) score below 19.
* Subjects must not have a previous Clinical Dementia Rating (CDR) global score of ≥2.
* Subjects must not have a Montreal Cognitive Assessment (MoCA)43 score of below 18 previously or during their screening evaluation.
* Subjects must not demonstrate a progression of aMCI to dementia at screening based on the best judgement of a study Clinical Neuropsychologist.
* Subjects must not currently participate in a high level of physical activity prior to study start as assessed by the International Physical Activity Questionnaire (IPAQ) at screening.
* Subjects must not endorse that they are unable to participate in moderate intensity aerobic activities, such as fast walking or passing/kicking a ball to a partner at screening.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bramen, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Pacific Brain Health Center, Santa Monica, California, United States

REFERENCES:
- [Background] Rozzini L, Chilovi BV, Conti M, Bertoletti E, Delrio I, Trabucchi M, Padovani A. Conversion of amnestic Mild Cognitive Impairment to dementia of Alzheimer type is independent to memory deterioration. Int J Geriatr Psychiatry. 2007 Dec;22(12):1217-22. doi: 10.1002/gps.1816. PMID 17562522
- [Background] Naismith SL, Glozier N, Burke D, Carter PE, Scott E, Hickie IB. Early intervention for cognitive decline: is there a role for multiple medical or behavioural interventions? Early Interv Psychiatry. 2009 Feb;3(1):19-27. doi: 10.1111/j.1751-7893.2008.00102.x. PMID 21352171
- [Background] Merrill DA, Small GW. Prevention in psychiatry: effects of healthy lifestyle on cognition. Psychiatr Clin North Am. 2011 Mar;34(1):249-61. doi: 10.1016/j.psc.2010.11.009. Epub 2010 Dec 16. PMID 21333851
- [Background] Rodakowski J, Saghafi E, Butters MA, Skidmore ER. Non-pharmacological interventions for adults with mild cognitive impairment and early stage dementia: An updated scoping review. Mol Aspects Med. 2015 Jun-Oct;43-44:38-53. doi: 10.1016/j.mam.2015.06.003. Epub 2015 Jun 10. PMID 26070444
- [Background] Smith PJ, Blumenthal JA, Hoffman BM, Cooper H, Strauman TA, Welsh-Bohmer K, Browndyke JN, Sherwood A. Aerobic exercise and neurocognitive performance: a meta-analytic review of randomized controlled trials. Psychosom Med. 2010 Apr;72(3):239-52. doi: 10.1097/PSY.0b013e3181d14633. Epub 2010 Mar 11. PMID 20223924
- [Background] Sofi F, Valecchi D, Bacci D, Abbate R, Gensini GF, Casini A, Macchi C. Physical activity and risk of cognitive decline: a meta-analysis of prospective studies. J Intern Med. 2011 Jan;269(1):107-17. doi: 10.1111/j.1365-2796.2010.02281.x. Epub 2010 Sep 10. PMID 20831630
- [Background] Huckans M, Hutson L, Twamley E, Jak A, Kaye J, Storzbach D. Efficacy of cognitive rehabilitation therapies for mild cognitive impairment (MCI) in older adults: working toward a theoretical model and evidence-based interventions. Neuropsychol Rev. 2013 Mar;23(1):63-80. doi: 10.1007/s11065-013-9230-9. Epub 2013 Mar 8. PMID 23471631
- [Background] Snowden M, Steinman L, Mochan K, Grodstein F, Prohaska TR, Thurman DJ, Brown DR, Laditka JN, Soares J, Zweiback DJ, Little D, Anderson LA. Effect of exercise on cognitive performance in community-dwelling older adults: review of intervention trials and recommendations for public health practice and research. J Am Geriatr Soc. 2011 Apr;59(4):704-16. doi: 10.1111/j.1532-5415.2011.03323.x. Epub 2011 Mar 25. PMID 21438861
- [Background] Kramer AF, Colcombe S. Fitness Effects on the Cognitive Function of Older Adults: A Meta-Analytic Study-Revisited. Perspect Psychol Sci. 2018 Mar;13(2):213-217. doi: 10.1177/1745691617707316. PMID 29592650
- [Background] Bamidis PD, Vivas AB, Styliadis C, Frantzidis C, Klados M, Schlee W, Siountas A, Papageorgiou SG. A review of physical and cognitive interventions in aging. Neurosci Biobehav Rev. 2014 Jul;44:206-20. doi: 10.1016/j.neubiorev.2014.03.019. Epub 2014 Apr 4. PMID 24705268
- [Background] Zhu X, Yin S, Lang M, He R, Li J. The more the better? A meta-analysis on effects of combined cognitive and physical intervention on cognition in healthy older adults. Ageing Res Rev. 2016 Nov;31:67-79. doi: 10.1016/j.arr.2016.07.003. Epub 2016 Jul 14. PMID 27423932
- [Background] Law LL, Barnett F, Yau MK, Gray MA. Effects of combined cognitive and exercise interventions on cognition in older adults with and without cognitive impairment: a systematic review. Ageing Res Rev. 2014 May;15:61-75. doi: 10.1016/j.arr.2014.02.008. Epub 2014 Mar 12. PMID 24632497
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] McEwen SC, Siddarth P, Rahi B, Kim Y, Mui W, Wu P, Emerson ND, Lee J, Greenberg S, Shelton T, Kaiser S, Small GW, Merrill DA. Simultaneous Aerobic Exercise and Memory Training Program in Older Adults with Subjective Memory Impairments. J Alzheimers Dis. 2018;62(2):795-806. doi: 10.3233/JAD-170846. PMID 29480182
- [Background] Black JE, Isaacs KR, Anderson BJ, Alcantara AA, Greenough WT. Learning causes synaptogenesis, whereas motor activity causes angiogenesis, in cerebellar cortex of adult rats. Proc Natl Acad Sci U S A. 1990 Jul;87(14):5568-72. doi: 10.1073/pnas.87.14.5568. PMID 1695380
- [Background] van Praag H, Christie BR, Sejnowski TJ, Gage FH. Running enhances neurogenesis, learning, and long-term potentiation in mice. Proc Natl Acad Sci U S A. 1999 Nov 9;96(23):13427-31. doi: 10.1073/pnas.96.23.13427. PMID 10557337
- [Background] Kleim JA, Markham JA, Vij K, Freese JL, Ballard DH, Greenough WT. Motor learning induces astrocytic hypertrophy in the cerebellar cortex. Behav Brain Res. 2007 Mar 28;178(2):244-9. doi: 10.1016/j.bbr.2006.12.022. Epub 2007 Jan 25. PMID 17257689
- [Background] Hotting K, Roder B. Beneficial effects of physical exercise on neuroplasticity and cognition. Neurosci Biobehav Rev. 2013 Nov;37(9 Pt B):2243-57. doi: 10.1016/j.neubiorev.2013.04.005. Epub 2013 Apr 25. PMID 23623982
- [Background] Lista I, Sorrentino G. Biological mechanisms of physical activity in preventing cognitive decline. Cell Mol Neurobiol. 2010 May;30(4):493-503. doi: 10.1007/s10571-009-9488-x. Epub 2009 Dec 30. PMID 20041290
- [Background] Novkovic T, Mittmann T, Manahan-Vaughan D. BDNF contributes to the facilitation of hippocampal synaptic plasticity and learning enabled by environmental enrichment. Hippocampus. 2015 Jan;25(1):1-15. doi: 10.1002/hipo.22342. Epub 2014 Aug 28. PMID 25112659
- [Background] Vaynman S, Ying Z, Gomez-Pinilla F. Exercise induces BDNF and synapsin I to specific hippocampal subfields. J Neurosci Res. 2004 May 1;76(3):356-62. doi: 10.1002/jnr.20077. PMID 15079864
- [Background] Gomez-Pinilla F, Vaynman S, Ying Z. Brain-derived neurotrophic factor functions as a metabotrophin to mediate the effects of exercise on cognition. Eur J Neurosci. 2008 Dec;28(11):2278-87. doi: 10.1111/j.1460-9568.2008.06524.x. PMID 19046371
- [Background] Neeper SA, Gomez-Pinilla F, Choi J, Cotman C. Exercise and brain neurotrophins. Nature. 1995 Jan 12;373(6510):109. doi: 10.1038/373109a0. No abstract available. PMID 7816089
- [Background] Gunstad J, Benitez A, Smith J, Glickman E, Spitznagel MB, Alexander T, Juvancic-Heltzel J, Murray L. Serum brain-derived neurotrophic factor is associated with cognitive function in healthy older adults. J Geriatr Psychiatry Neurol. 2008 Sep;21(3):166-70. doi: 10.1177/0891988708316860. Epub 2008 May 23. PMID 18503034
- [Background] Erickson KI, Miller DL, Roecklein KA. The aging hippocampus: interactions between exercise, depression, and BDNF. Neuroscientist. 2012 Feb;18(1):82-97. doi: 10.1177/1073858410397054. Epub 2011 Apr 29. PMID 21531985
- [Background] Nascimento CM, Pereira JR, de Andrade LP, Garuffi M, Talib LL, Forlenza OV, Cancela JM, Cominetti MR, Stella F. Physical exercise in MCI elderly promotes reduction of pro-inflammatory cytokines and improvements on cognition and BDNF peripheral levels. Curr Alzheimer Res. 2014;11(8):799-805. doi: 10.2174/156720501108140910122849. PMID 25212919
- [Background] McMorris T, Davranche K, Jones G, Hall B, Corbett J, Minter C. Acute incremental exercise, performance of a central executive task, and sympathoadrenal system and hypothalamic-pituitary-adrenal axis activity. Int J Psychophysiol. 2009 Sep;73(3):334-40. doi: 10.1016/j.ijpsycho.2009.05.004. Epub 2009 May 18. PMID 19454298
- [Background] Grudzien A, Shaw P, Weintraub S, Bigio E, Mash DC, Mesulam MM. Locus coeruleus neurofibrillary degeneration in aging, mild cognitive impairment and early Alzheimer's disease. Neurobiol Aging. 2007 Mar;28(3):327-35. doi: 10.1016/j.neurobiolaging.2006.02.007. Epub 2006 Mar 29. PMID 16574280
- [Background] Klimesch W, Sauseng P, Hanslmayr S. EEG alpha oscillations: the inhibition-timing hypothesis. Brain Res Rev. 2007 Jan;53(1):63-88. doi: 10.1016/j.brainresrev.2006.06.003. Epub 2006 Aug 1. PMID 16887192
- [Background] Richard Clark C, Veltmeyer MD, Hamilton RJ, Simms E, Paul R, Hermens D, Gordon E. Spontaneous alpha peak frequency predicts working memory performance across the age span. Int J Psychophysiol. 2004 Jun;53(1):1-9. doi: 10.1016/j.ijpsycho.2003.12.011. PMID 15172130
- [Background] Vlahou EL, Thurm F, Kolassa IT, Schlee W. Resting-state slow wave power, healthy aging and cognitive performance. Sci Rep. 2014 May 29;4:5101. doi: 10.1038/srep05101. PMID 24869503
- [Background] Klimesch W. EEG alpha and theta oscillations reflect cognitive and memory performance: a review and analysis. Brain Res Brain Res Rev. 1999 Apr;29(2-3):169-95. doi: 10.1016/s0165-0173(98)00056-3. PMID 10209231
- [Background] Li Y, Zhao Z, Cai J, Gu B, Lv Y, Zhao L. The Frequency-Dependent Aerobic Exercise Effects of Hypothalamic GABAergic Expression and Cardiovascular Functions in Aged Rats. Front Aging Neurosci. 2017 Jun 30;9:212. doi: 10.3389/fnagi.2017.00212. eCollection 2017. PMID 28713263
- [Background] Bondi MW, Edmonds EC, Jak AJ, Clark LR, Delano-Wood L, McDonald CR, Nation DA, Libon DJ, Au R, Galasko D, Salmon DP. Neuropsychological criteria for mild cognitive impairment improves diagnostic precision, biomarker associations, and progression rates. J Alzheimers Dis. 2014;42(1):275-89. doi: 10.3233/JAD-140276. PMID 24844687
- [Background] Bondi MW, Jak AJ, Delano-Wood L, Jacobson MW, Delis DC, Salmon DP. Neuropsychological contributions to the early identification of Alzheimer's disease. Neuropsychol Rev. 2008 Mar;18(1):73-90. doi: 10.1007/s11065-008-9054-1. Epub 2008 Mar 18. PMID 18347989
- [Background] Clark LR, Delano-Wood L, Libon DJ, McDonald CR, Nation DA, Bangen KJ, Jak AJ, Au R, Salmon DP, Bondi MW. Are empirically-derived subtypes of mild cognitive impairment consistent with conventional subtypes? J Int Neuropsychol Soc. 2013 Jul;19(6):635-45. doi: 10.1017/S1355617713000313. Epub 2013 Apr 3. PMID 23552486
- [Background] Edmonds EC, Delano-Wood L, Clark LR, Jak AJ, Nation DA, McDonald CR, Libon DJ, Au R, Galasko D, Salmon DP, Bondi MW; Alzheimer's Disease Neuroimaging Initiative. Susceptibility of the conventional criteria for mild cognitive impairment to false-positive diagnostic errors. Alzheimers Dement. 2015 Apr;11(4):415-24. doi: 10.1016/j.jalz.2014.03.005. Epub 2014 May 22. PMID 24857234
- [Background] Nuriel T, Angulo SL, Khan U, Ashok A, Chen Q, Figueroa HY, Emrani S, Liu L, Herman M, Barrett G, Savage V, Buitrago L, Cepeda-Prado E, Fung C, Goldberg E, Gross SS, Hussaini SA, Moreno H, Small SA, Duff KE. Neuronal hyperactivity due to loss of inhibitory tone in APOE4 mice lacking Alzheimer's disease-like pathology. Nat Commun. 2017 Nov 13;8(1):1464. doi: 10.1038/s41467-017-01444-0. PMID 29133888
- [Background] Jak AJ, Bondi MW, Delano-Wood L, Wierenga C, Corey-Bloom J, Salmon DP, Delis DC. Quantification of five neuropsychological approaches to defining mild cognitive impairment. Am J Geriatr Psychiatry. 2009 May;17(5):368-75. doi: 10.1097/JGP.0b013e31819431d5. PMID 19390294
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Miller KJ, Siddarth P, Gaines JM, Parrish JM, Ercoli LM, Marx K, Ronch J, Pilgram B, Burke K, Barczak N, Babcock B, Small GW. The memory fitness program: cognitive effects of a healthy aging intervention. Am J Geriatr Psychiatry. 2012 Jun;20(6):514-23. doi: 10.1097/JGP.0b013e318227f821. PMID 21765343
- [Background] Colcombe SJ, Erickson KI, Raz N, Webb AG, Cohen NJ, McAuley E, Kramer AF. Aerobic fitness reduces brain tissue loss in aging humans. J Gerontol A Biol Sci Med Sci. 2003 Feb;58(2):176-80. doi: 10.1093/gerona/58.2.m176. PMID 12586857
- [Background] Foster C, Jackson AS, Pollock ML, Taylor MM, Hare J, Sennett SM, Rod JL, Sarwar M, Schmidt DH. Generalized equations for predicting functional capacity from treadmill performance. Am Heart J. 1984 Jun;107(6):1229-34. doi: 10.1016/0002-8703(84)90282-5. No abstract available. PMID 6720550
- [Background] Polacchini A, Metelli G, Francavilla R, Baj G, Florean M, Mascaretti LG, Tongiorgi E. A method for reproducible measurements of serum BDNF: comparison of the performance of six commercial assays. Sci Rep. 2015 Dec 10;5:17989. doi: 10.1038/srep17989. PMID 26656852
- [Background] Segal SK, Cotman CW, Cahill LF. Exercise-induced noradrenergic activation enhances memory consolidation in both normal aging and patients with amnestic mild cognitive impairment. J Alzheimers Dis. 2012;32(4):1011-8. doi: 10.3233/JAD-2012-121078. PMID 22914593
- [Background] Will PM, Walter JD. Exercise testing: improving performance with a ramped Bruce protocol. Am Heart J. 1999 Dec;138(6 Pt 1):1033-7. doi: 10.1016/s0002-8703(99)70067-0. PMID 10577432
- [Background] Balady GJ, Chaitman B, Driscoll D, Foster C, Froelicher E, Gordon N, Pate R, Rippe J, Bazzarre T. Recommendations for cardiovascular screening, staffing, and emergency policies at health/fitness facilities. Circulation. 1998 Jun 9;97(22):2283-93. doi: 10.1161/01.cir.97.22.2283. No abstract available. PMID 9631884
- [Background] Gualtieri CT, Johnson LG. Reliability and validity of a computerized neurocognitive test battery, CNS Vital Signs. Arch Clin Neuropsychol. 2006 Oct;21(7):623-43. doi: 10.1016/j.acn.2006.05.007. Epub 2006 Oct 2. PMID 17014981
- See also: World Health Organization (WHO) definitions — http://www.who.int/mediacentre/factsheets/fs362/en/
- See also: Rivermead Behavioural Memory Test - Third Edition (RBMT-3) — https://www.pearsonclinical.co.uk/Psychology/AdultCognitionNeuropsychologyandLanguage/AdultMemory/RivermeadBehaviouralMemoryTestThirdEditionRBMT3/RivermeadBehaviouralMemoryTestThirdEditionRBMT3.aspx
- See also: Use of the Functional Activities Questionnaire in Older Adults with Dementia — https://www.alz.org/careplanning/downloads/functional-activities-questionnaire.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 22 participants that were consented, 1 failed screening due to MoCa score and 2 were lost to follow up. Participants were then screened prior to randomization, which included exercise clearance and full neurocognitive assessment. Of the 19 that were screened, 12 were randomized because 6 failed to meet criteria due to neurocognitive assessment, and 1 was unable to obtain clearance to participate in an exercise intervention.
Period: Overall Study
Arm/Group | Group 1 (No Treatment) | Group 2 (Experimental)
Started | 4 | 8
Completed | 3 | 2
Not Completed | 1 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (No Treatment) | Group 2 (Experimental) | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (6.4) | 69.7 (4.5) | 71.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Memory Function Composite Score
Description: Global Z-Score including results from RAVLT (Rey's Auditory Verbal Learning Test), Wechsler Memory Scale Fourth Edition (WMS-IV) Logical Memory and Visual Reproduction tests.
  The global z score was constructed by:
  First z-transforming all raw test scores (RAVLT, Logical Memory (LM) I Total, LM II Total, Visual Reproduction (VR) I and VR II) Averaging over RAVLT Z, LM Z, and VR Z to obtain a global Z 0=sample mean; higher scores indicate better outcomes.
Time Frame: Baseline, approximately 3 months and approximately 6 months
Population: Of the 8 participants that were randomized into the intervention, only 7 participated in baseline assessments. Of the 7 with baseline data, only 2 completed follow up assessments.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Group 1 (No Treatment) | Group 2 (Experimental)
Number analyzed (Participants) | 3 | 7
Z-score
  Baseline | 0.5 (0.84) | -0.21 (1.80)
  3 Months: number analyzed (Participants) | 3 | 2
  3 Months | 0.87 (0.49) | -1.30 (4.19)
  6 Months: number analyzed (Participants) | 3 | 2
  6 Months | 0.66 (1.63) | -0.98 (4.33)

2. Primary Outcome: Functional Abilities
Description: Assessed using the Multifactorial Memory Questionnaire (MMQ) Satisfaction Sub-scale (0-72 points). Higher scores indicate better outcomes.
Time Frame: Baseline, approximately 3 months and approximately 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 (No Treatment) | Group 2 (Experimental)
Number analyzed (Participants) | 3 | 7
scores on a scale
  Baseline | 24.67 (13.01) | 26.86 (15.65)
  3 Months: number analyzed (Participants) | 3 | 2
  3 Months | 26.33 (14.19) | 19.00 (11.31)
  6 Months: number analyzed (Participants) | 3 | 2
  6 Months | 32.67 (16.77) | 21.00 (5.66)

3. Secondary Outcome: Resting Brain-derived Neurotrophic Factor (BDNF)
Description: Resting level of serum-derived BDNF
Time Frame: Baseline and approximately 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Resting Norepinephrine (NE)
Description: Resting level of plasma-derived norepinephrine (NE)
Time Frame: Baseline and approximately 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Group 1 (No Treatment) | Group 2 (Experimental)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 3/4 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (No Treatment) (N=4) | Group 2 (Experimental) (N=8)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Acute sprain of ligament of neck due to car accident. Not related to intervention.
Rib pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Contusion due to a car accident. Not related to intervention.
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Possible concussion due to car accident. Not related to the intervention.
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (General disorders) | 1 (1) | 0 (0) — Back surgery from pre-existing condition. Not related to intervention
Tooth pain (Infections and infestations) | 1 (1) | 0 (0) — Root canal. Not related to the intervention.
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Not related to the intervention
Limb pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Avulsion of skin of left forearm and contusion of left upper arm, due to car accident, due to car accident. Not related to intervention.
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not due to intervention
Shingles (Infections and infestations) | 1 (1) | 0 (0) — Not due the intervention.

LIMITATIONS AND CAVEATS:
Early termination due to small number of participants recruited and low intervention completion rates led to small numbers of subjects analyzed. One of the participants that completed the study in the intervention arm had a mid-trial concussion. Data are not interpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04185298/Prot_SAP_000.pdf